CLINICAL TRIAL: NCT05714111
Title: Radiology Registry on Pancreatic Malignancies
Acronym: RadonPams
Status: Recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Francesco De Cobelli, Head of Radiology, IRCCS San Raffaele
Other Study IDs: RadonPams
Record Dates: First submitted 2023-01-25; First posted 2023-02-06 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Pancreatic Cancer; Pancreas Neoplasm; Pancreas Disease; Pancreas Cyst
MeSH Terms: conditions — Pancreatic Neoplasms; Pancreatic Diseases; Pancreatic Cyst | interventions — Methods

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Biopsy or intraoperatory samples according to standard of care
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Radiology evaluations and interventions — Diagnostic and interventional radiology procedures

SUMMARY:
The purpose of this study is to collect all radiological data which evaluated with clinical data may help assess malignancy and prognosis of pancreatic disease.This registry aims to collect retrospective data from 2014 and prospective data until 2027 with a maximum follow-up of 3 years per patient.

DETAILED DESCRIPTION:
Single center, observational (retrospective and prospective) will collect all available parameters to assess the clinical outcome of the patients (progression free survival (PFS), overall survival (OS), local progression free survival LTPFS), response to treatment) with pancreatic neoplasms presenting to San Raffaele. Patient assignment to a given diagnostic and/or therapeutic procedure is not related to random assignment methods but is part of the ordinary therapeutic strategy planned for each patient on an individual basis and after multidisciplinary discussion.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* Patients with suspect (planned for investigation) or diagnosed pancreatic cancer at any stage.
* able and willing to sign informed consent

Exclusion Criteria:

* Patients with non-primary pancreatic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with pancreatic adenocarcinoma, pancreatic neuroendocrine tumors, rare forms of pancreatic cancer (such as ampullary cancer, adenosquamous carcinomas, squamous cell carcinomas, signet ring cell carcinomas, undifferentiated carcinomas, and undifferentiated carcinomas with giant cells) and cystic neoplasms.
Sampling Method: Non-Probability Sample
Enrollment: 1300 (Estimated)
Dates: Start 2022-03-04 (Actual); Primary Completion 2027-03-30 (Estimated); Study Completion 2030-03-30 (Estimated)

PRIMARY OUTCOMES:
Progression- free survival | From date of intervention until the date of first documented progression, up to a maximum of 3 years
  Time from start of observation to disease progression
Local progression free survival | From date of intervention until the date of first documented local progression assessed up to a maximum of 3 years
  Time between (start of) a locoregional treatment and local disease progression

SECONDARY OUTCOMES:
Overall Survival | From date of treatment until the date of death from any cause assessed up to 3 years
  The length of time from either the date of diagnosis or the start of treatment for a disease, in which the patients are still alive

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Radiology, IRCCS Ospedale San Raffaele, Milan, Italy